CLINICAL TRIAL: NCT03323424
Title: Phase II Trial Assessing the Efficacy of Immuno-Radiation Abscopal Effect in Patients With Metastatic Cancers (IRAM)
Brief Title: Phase II Trial Assessing the Efficacy of Immuno-Radiation Abscopal Effect in Patients With Metastatic Cancers
Acronym: IRAM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patient enrolled during the authorized period
Sponsor: Institut de Cancérologie de la Loire (Other)
Collaborators: Saint-Louis Hospital, Paris, France (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0301; 2017-A02043-50 (Other: ANSM)
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Breast Cancer; Metastatic Colorectal Cancer; Metastatic Head and Neck Cancer
Keywords: Metastatic cancer; Abscopal effect; Ionizing radiation; Antibody-Dependant Cell Cytotoxicity (ADCC); Immuno-Radiation effect; Stereotactic Body Radio-Therapy (SBRT); Targeted therapies
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Neoplasm Metastasis | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic treatment + Stereotactic Body Radio-Therapy (SBRT) (Experimental): Patients with metastatic breast, colorectal or head or neck cancers and corresponding with the inclusion criteria will receive a systemic treatment, according to the usual practice, but also a Stereotactic Body Radio-Therapy (SBRT).
  Interventions: Radiation: Systemic treatment + Stereotactic Body Radio-Therapy (SBRT)
- Systemic treatment (Active Comparator): Patients with metastatic breast, colorectal or head or neck cancers and corresponding with the inclusion criteria will receive a systemic treatment, according to the usual practice.
  Interventions: Other: Systemic treatment

INTERVENTIONS:
Radiation: Systemic treatment + Stereotactic Body Radio-Therapy (SBRT) — According to the usual practice, patients will receive their systemic treatment, composed of :
  * Taxane + trastuzumab +pertuzumab for metastatic breast cancers;
  * FOLFOX or FOLFIRI + cetuximab for metastatic colorectal cancers;
  * 5FU-Platine + cetuximab for metastatic head and neck cancers; for six cycles and a maintenance of the targeted therapy until progression or unacceptable toxicity.
  If progression occurs before the 6th cycles, patients could receive a different line of treatment, according to the usual practice.
  In addition to the systemic treatment, patients randomized into this experimental group will receive a SBRT of 45Gy in 3 fractions for hepatic and pulmonary metastasis, 27Gy in 3 fractions for bone metastasis and 33 Gy in 3 fractions for intra-cranial metastasis.
  Arms: Systemic treatment + Stereotactic Body Radio-Therapy (SBRT)
Other: Systemic treatment — According to the usual practice, patients will receive their systemic treatment, composed of :
  * Taxane + trastuzumab +pertuzumab for metastatic breast cancers;
  * FOLFOX or FOLFIRI + cetuximab for metastatic colorectal cancers;
  * 5FU-Platine + cetuximab for metastatic head and neck cancers; for six cycles and a maintenance of the targeted therapy until progression or unacceptable toxicity.
  If progression occurs before the 6th cycles, patients could receive a different line of treatment, according to the usual practice.
  Arms: Systemic treatment

SUMMARY:
The proposed theory is based on combination of radiation therapy with usual targeted therapies capable of ADCC (Antibody-Dependant Cell Cytotoxicity). This association could enhance in a additive/synergistic way the benefic impact of immune system activation on tumor control. Stereotactic Body Radio-Therapy (SBRT) will be combined with the first line chemotherapy for metastatic breast, colorectal or VADS (upper aerodigestive tract) cancers. The IRAM study objective is to highlight a possible abscopal effect of this combination for metastatic cancer patients.

DETAILED DESCRIPTION:
Nowadays, metastatic cancer treatment is evolving with systemic treatments (target therapies and immunotherapies). Combinations and new therapeutic schemes have recently boosted the interest for an effect called "abscopal". This effect is based on the immune-stimulating effect of high doses ionizing radiations, but also on synergistic association with systemic treatment with immunologic mechanisms. This effect could enhance the tumor local control, but also its distant control.

Numerous preclinical evidences as well as some clinical case reports described the abscopal effect.

Ongoing clinical studies are investigating with radiotherapy abscopal effect alone, or associated with immunotherapies (anti-CTLA-4, PD-1 or PDL-1). The present study proposes a new association, based on an original biological rational. The proposed theory is based on combination of radiation therapy with usual targeted therapies capable of ADCC (Antibody-Dependant Cell Cytotoxicity). This association could enhance in an additive/synergistic way the benefic impact of immune system activation on tumor control.

In the present study, Stereotactic Body Radio-Therapy (SBRT) will be combined to the standard systemic treatment for first line treatment of metastatic breast, colorectal and VADS (upper aerodigestive tract) cancers. Indeed, these treatments have in common the use of target therapies capable of ADCC.

The IRAM study objective is to highlight a possible abscopal effect of this combination for metastatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a metastatic breast adenocarcinoma HER2+, a metastatic squamous carcinoma of VADS, or a colorectal adenocarcinoma with a wild status for RAS (NRAS and KRAS)
* Patient presenting at least two measurable metastases (according to the RECIST v1.1 criteria):
* At least one eligible to SBRT (hepatic, pulmonary, bone or intra-cranial metastasis, with a diameter between 1 and 4cm)
* At least one non irradiated measurable metastasis
* Performance Status corresponding to 0, 1, or 2
* Realisation of a PET (Positron Emission Tomography)-Scanner and a TAP (Thoraco-AbdominoPelvic)-Scanner 30 days maximum before inclusion
* Informed consent patient
* Patients affiliated to a social security scheme.

Exclusion Criteria:

* Patient presenting a known non-indication or contraindication to the first line treatment administered
* Pregnant or nursing women
* Patient with an another cancer during the 5 last years, excepting basocellular carcinoma, and skin epidermoid carcinoma
* Patient presenting a non-controlled pain linked to the cancer
* Patient presenting a non-controlled hypercalcemia or symptomatic hypercalcemia needing an ongoing use of bisphosphonates or denosumab.
* Patient presenting an inflammatory pathology or active autoimmune pathology or history of.
* Patient having received one or more vaccines during the 4 weeks preceding the beginning of the systemic treatment.
* Patient currently using corticosteroids or other immune-suppressors during the two weeks before inclusion, and any other situation where this kind of treatments could be necessary during the study.
* Patient deprive of liberty or under administrative supervision, patients with an impossible take care supervision for psychological or geographical reasons.
* Stereotactic Body Radio-Therapy (SBRT) must not include metastases localized in the 3 centimeters of the structure previously irradiated.
* Patient presenting serious active comorbidities defined by the protocol.
* Known seropositivity to the HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate without progression for patients with metastatic breast cancer | 18 months
  The rate of survival without progression according to the RECIST (v1.1) criteria for patients with metastatic breast cancer will be calculated at 18 months after the beginning of the systemic treatment.
Survival rate without progression for metastatic head and neck cancer | 6 months
  The rate of survival without progression according to the RECIST (v1.1) criteria for patients with head and neck cancer will be calculated at 6 months after the beginning of the systemic treatment.
Survival rate without progression for patients with metastatic colorectal cancer | 9 months
  The rate of survival without progression according to the RECIST (v1.1) criteria for patients with colorectal cancer will be calculated at 9 months after the beginning of the systemic treatment.

SECONDARY OUTCOMES:
Response rate on predetermined metastatic abscopal sites | 3 months
  The response rate on predetermined metastatic abscopal sites will be evaluated at 3 months after the beginning of the systemic treatment according to the RECIST v1.1 criteria.
Response rate on the irradiated site | 3 months
  The response rate on the irradiated site will be evaluated at 3 months after the beginning of the systemic treatment according to the RECIST v1.1 criteria.
Progression-free survival (PFS) | 5 years
  The median PFS according to the RECIST v1.1 criteria will be reported at 5 years after the beginning of the systemic treatment.
Overall survival (OS) | 5 years
  The OS will be reported at 5 years after the beginning of the systemic treatment.
Toxicity of the treatments combination | 6 cycles
  During the first line of systemic treatment (six cycles of treatment maximum), the number and the grade (CTCAE v4.4) of toxicities related to the systemic treatment /Radiation therapy combination will be reported.
Toxicity of the treatments combination | 5 years
  Sub-group analysis will be performed following the 3 binary stratification criteria: total number of metastasis, localization of the irradiated metastasis and irradiated volume.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Magné, PhD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (6):
- France (6):
  - Clinique Claude Bernard, Albi
  - Centre Léonard de Vinci, Dechy
  - Centre Hospitalier Privé Saint Gregoire, Saint-Grégoire
  - CHU de St-Etienne, Saint-Priest-en-Jarez
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Marie Curie, Valence

IPD SHARING:
Plan to Share IPD: No